CLINICAL TRIAL: NCT06617390
Title: Real-world Treatment Patterns and Outcomes in Chinese Advanced NSCLC Patients Who Previously Received at Least 2 Line Treatment: a Multi-center, Non-interventional and Retrospective Real-world Study (RECAP)
Brief Title: A Study of Real-world Treatment Patterns and Outcomes in Chinese Advanced NSCLC Patients Who Previously Received at Least 2 Line Treatments
Acronym: RECAP
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS1062-0001-NIS-MA
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AGA Cohort: NSCLC participants with AGA that received second-line or above therapies treatment.
  Interventions: Other: No drug
- Non-AGA Cohort: NSCLC participants with non-AGA that received second-line or above therapies treatment.
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — This is a non-interventional study and no study drug will be provided.

SUMMARY:
This study will retrospectively collect data of patients with advanced non-small cell lung cancer who have received at least 2 line treatment to investigate treatment patterns, relevant outcomes, and biomarkers detection patterns in Chinese patients with Actionable Genomic Alterations (AGA) or non-AGA.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged ≥18 years when diagnosed with advanced NSCLC.
2. Histologically or cytologically confirmed stage IV NSCLC.
3. For non-AGA participants , second- or third-line systemic treatment occurred between September 1, 2019 and December 31, 2022, and participants received corresponding immunotherapy in the first or second line.
4. For AGA participants , second- or third-line systemic treatment occurred between September 1, 2019 and December 31, 2022. Among them, participants with documented positive result for EGFR, ALK, or ROS1 testing received corresponding targeted therapy in the first or second line.

Exclusion Criteria:

This study excludes participants who met any of the following criteria.

1. Having records of participation or past participation in clinical trial for lung cancer within the data collection period of the study.
2. Participants with a concomitant cancer at the time of diagnosis of NSCLC (except for non-metastatic non-melanoma skin cancers, in situ or benign neoplasms). Occurrence of cancer within 5 years after NSCLC diagnosis will be considered as secondary cancer.
3. Histology of the tumor is small cell lung cancer, neuroendocrine in origin, or a mixed histologic type with small cell and non-small cell lung cancers.
4. Participants with significantly missing medical record data or patients deemed inappropriate for inclusion by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced NSCLC who have received at least 2L treatment between September 1, 2019, and December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 1041 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Percentage of real-world treatment regimens for second- or third-line therapy in patients with advanced NSCLC | 40 months

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Cancer Hospital, Beijing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Affiliated Hospital of Soochow University, Suzhou

IPD SHARING:
Plan to Share IPD: No